CLINICAL TRIAL: NCT06726005
Title: Impact of Functional Appliances on 3D Craniodentofacial Characteristics and Reported Sleep Related Breathing Disorders in Children
Brief Title: 3D Characteristics, Functional Appliances and Sleep Related Breathing Disorders
Acronym: FA PSQ HR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Visnja Katic, Associate Professor, University of Rijeka
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: uniri-iskusni-biomed-23-36
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-04

CONDITIONS: Retrognathic Mandible
Keywords: PSQ; Twin block; 3D facial scan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Functional appliance group (Experimental): Upon diagnostics, functional appliance Twin block will be proposed to the participants for one year.
  Interventions: Device: functional appliance twin block

INTERVENTIONS:
Device: functional appliance twin block — 3D facial scans will be taken (prior to the treatment, at rest and at mandible moved forward to class I dental relation (Fraenkel manouver)) and at the end of treatment, one year later.

SUMMARY:
Facial scans of the patients eligible for the functional appliance treatment (Twin Block appliance) will be taken prior to and after the end of treatment. Also, a facial scan of the predicted final outcome will be taken, and compared to the actual final outcome. Parents / caregivers will fill out the Pediatric Sleep Questionnaire (PSQ) prior to and upon the end of treatment to asses perceived influence on sleep related breathing problems in their children.

DETAILED DESCRIPTION:
The harmonious growth of the upper and lower jaw enables further favorable development of the orofacial region and the functions of breathing, chewing, swallowing and speaking, as well as the general growth and development of the child. Translation into Croatian and administration of the questionnaire for early detection of sleep disorders related to breathing in children (PSQ) will enable triage and early recognition of children with sleep disorders, which also affect general psycho-physical development. The impact of functional appliance therapy (FA) on changes in craniodentofacial characteristics, dimensions of the upper airway and sleep problems in children will be determined. The non-invasive three-dimensional representation of the face surface provides information about the surface and volume of the observed object, which is used for better diagnostics and therapy planning. Class II is a frequent malocclusion, characterized by a discrepancy of sagittal interjaw relationships. The diagnostic method, which helps in deciding on a therapeutic approach, is the so-called Fränkel maneuver (FM). By comparing the observation of the soft tissue profile of the subjects at rest and after the application of FM, a decision is made on the therapeutic approach. Previous research indicates the validity of using FM in making a decision about FN therapy, with high reliability and consistency. The analysis of latero-lateral (LL) X-ray cephalograms in numerous studies has provided a series of data, which is used, among other things, to assess the remaining growth in order to apply FN therapy in a timely manner, but also to expect a desirable response. The evaluation of the success of therapy based on FM don't exist, because a reliable 2D analysis through LL cephalogram would require additional radiation of the subjects. Research indicates that the analysis of scan surfaces is more appropriate than the analysis of anatomical points for detection of the area and amount of changes.

ELIGIBILITY:
Inclusion Criteria:

* retrognathic mandible, increased overjet

Exclusion Criteria:

* craniodentofacial deformities

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Facial scan | from enrollment and predicted outcome to the end of treatment at one year on average
  Using stereophotographic camera, 3D facial scans will be taken, and superimposed to observe differences prior to and at the end of treatment. Also, predicted outcome (facial scan taken in Fraenkel manouver position (at start)) will be compared to the actual outcome after one year of treatment with functional appliance Twin Block.
PSQ questionnaire | from enrollment to the end of treatment at one year on average
  Parents / caregivers will fill out the PSQ questionnaire to assess influence of the functional appliance treatment on the sleep related breathing problems in their children.

SECONDARY OUTCOMES:
Latero-lateral cephalogram | from enrollment to the end of treatment at one year on average
  Cranio-dento-facial characteristics will be assessed prior to and at the end of treatment with functional appliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Rijeka, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
Data contain identifiable biometric data, and will be disclosed only upon reasonable request.